CLINICAL TRIAL: NCT07017036
Title: An Open- Label, Multicentre, Phase III Clinical Comparative Study to Evaluate the Efficacy, Safety and Pharmacokinetic Properties of Human Normal Immunoglobulin in Patients With Primary Immunodeficiency Disease
Brief Title: Efficacy, Safety and Pharmacokinetic of Virchow IVIG in PID Patients
Acronym: VBPL-IVIGP3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Virchow Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VBIVIG/2024-CT1; VBIVIG/2024-CT1 (Other: Virchow Biotech Private Ltd)
Record Dates: First submitted 2025-05-10; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Primary Immunodeficiency Diseases (PID)
Keywords: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Intervention Model Description: Treatment - Randomized - parallel group study
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm (Experimental): 200-800 mg/kg dose as a single infusion every 3 or 4 weeks. Patients will be treated with V-Immune from Week 0 (first dose) till Week 48 at an investigator-recommended dose.
  Interventions: Drug: IVIG-VImmune
- Reference (Active Comparator): Immuglo will be administered at 200-800 mg/kg dose as a single infusion every 3 or 4 weeks. Patients will be treated with V-Immune from Week 0 (first dose) till Week 48 at an investigator-recommended dose
  Interventions: Drug: IVIG-Immuglo

INTERVENTIONS:
Drug: IVIG-VImmune — V-Immune will be administered at 200-800 mg/kg dose as a single infusion every 3 or 4 weeks. Patients will be treated with V-Immune from Week 0 (first dose) till Week 48 at an investigator-recommended dose
  Arms: Test Arm
Drug: IVIG-Immuglo — Immuglo will be administered at 200-800 mg/kg dose as a single infusion every 3 or 4 weeks. Patients will be treated with V-Immune from Week 0 (first dose) till Week 48 at an investigator-recommended dose
  Arms: Reference

SUMMARY:
The study duration for individual patients will be up to 55 weeks for the 4-weekly and 3- weekly schedule of the treatment which includes 3 weeks for screening, 48 weeks for Study Medication administration and 4 weeks for follow-up assessments

DETAILED DESCRIPTION:
Eligible subjects will receive either test or reference as per the randomization in 1:1 ratio.

Test group: V-Immune will be administered at 200-800 mg/kg dose as a single infusion every 3 or 4 weeks. Patients will be treated with V-Immune from Week 0 (first dose) till Week 48 at an investigator-recommended dose.

Reference group: Immuglo will be administered at 200-800 mg/kg dose as a single infusion every 3 or 4 weeks. Patients will be treated with V-Immune from Week 0 (first dose) till Week 48 at an investigator-recommended dose

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 2 to 65 years.
2. Patients with confirmed diagnosis of primary immunodeficiency, predominantly antibody deficient, or common variable immunodeficiency (CVID) with a history of hypogammaglobulinemia (i.e., IgG<500 mg/dl) or X-linked agammaglobulinemia (XLA).
3. Treatment naive patients eligible to receive intravenous immunoglobulin or, patients already on intravenous immunoglobulin infusions every 3 or every 4 weeks for ≥6 months at a dose aimed to be between 200 and 800 mg/kg with at least two documented IgG trough levels in the previous two infusions before enrolment in the study.
4. The screening laboratory tests must meet the following criteria:

   1. WBC ≥3.5 x 109/L
   2. Neutrophils ≥1.5 x 109/L
   3. Platelets ≥100 x 109/L
   4. Serum transaminase ≤2 times the upper limit of normal
   5. Alkaline phosphatase levels ≤2 times the upper limit of normal
   6. Serum creatinine ≤150 µmol/L (≤1.7mg/dl)
5. Patients must be able to adhere to the study visit schedule and other protocol requirements.
6. If subject is a female and is

   a. -of child bearing potential, she should be practicing an acceptable method of birth control for the duration of tl1e study as suggested by the investigator, such as a combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier method), intrauterine device (IUD), or abstinence OR surgically sterile, bilateral tubal ligation done at least 6 months before the study should be documented
7. Patients/LAR must be capable of giving informed consent, and written consent must have been obtained prior to any study procedures.

Exclusion Criteria:

1. Pregnant women, nursing mothers or a planned pregnancy within 18 months of participation.
2. Patients requires any blood transfusion during the study.
3. Patients with T-cell related Severe combined immunodeficiency.
4. Patients with secondary immunodeficiency diseases
5. History or presence of any form of cancer prior to enrollment.
6. History of any autoimmune disease
7. Positive at screening for any markers of infectious blood borne viruses
8. History of adverse or allergic reactions to other IgG or blood products
9. Patients with selective IgA deficiency or antibodies IgA
10. History of acute renal failure or severe renal impairment, or deep venous thrombosis which in the opinion of the Investigator, may place the patient at unacceptable risk for study participation and may prevent the patient from completing the study.
11. History of congestive heart failure [New York Heart Association class III/IV] or unstable angina
12. Recent history of migraine, hyperprolinemia, and lymphoid malignancy.
13. Requirement for use of glucocorticosteroids above 0.15 mg of prednisone equivalent/kg/day and other immunosupressive drugs as concomitant medication.
14. History or presence of any medical or psychiatric condition or disease, or laboratory abnormality that, in the opinion of the Investigator, may place the patient at unacceptable risk for study participation and may prevent the patient from completing the study.
15. Participation in any clinical study within the previous 3 months
16. Patient, who in the opinion of the Investigator, is not suitable for participation in the clinical study

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary - Incidence of acute serious bacterial infections | 52 weeks
  incidence of acute serious bacterial infections per patient will be assessed at 52 weeks

SECONDARY OUTCOMES:
Secondary - Pharmacokinetics | 52 weeks
  To assess the Ig serum concentration - Cmax
Secondary Pharmacokinetics | 52 weeks
  To assess the IgG serum concentration Tmax
Safety of IVIG | 52 weeks
  Safety will be assessed

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - All India Institute of Medical Sciences, Nagpur, Maharashtra
  - Jyoti Nursing Home (P) Ltd., Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: No